CLINICAL TRIAL: NCT00003490
Title: Phase II to Treat Multiple Myeloma Patients With Cytoxan and Vincristine After Cycling Myeloma Cells With rHuGM-CSF
Brief Title: Combination Chemotherapy Following GM-CSF in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066529; CCF-IRB-1863; IMMUNEX-001.0743; NCI-V98-1458
Record Dates: First submitted 1999-11-01; First posted 2004-05-21 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2001-03

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — sargramostim; Cyclophosphamide; Prednisone; Vincristine

INTERVENTIONS:
Biological: sargramostim
Drug: cyclophosphamide
Drug: prednisone
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. GM-CSF may make cancer cells more sensitive to the effects of chemotherapy. Combining more than one drug with GM-CSF may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy, consisting of cyclophosphamide plus vincristine, following GM-CSF in treating patients with multiple myeloma that has not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate of multiple myeloma patients when treated with cyclophosphamide and vincristine after cycling myeloma cells with sargramostim (GM-CSF). II. Evaluate whether Labelling Index (LI) changes influenced by GM-CSF would predict a group of patients that will respond to this particular course specific design. III. Determine the toxicity of GM-CSF in these patients.

OUTLINE: Patients receive subcutaneous injections of sargramostim (GM-CSF) once a day for 5 days. Two to 3 days later, patients receive cyclophosphamide IV over 30-45 minutes on day 1, vincristine IV bolus on day 8, and oral prednisone 4 times a day on days 1-4. Patients also receive subcutaneous injections of GM-CSF starting on day 2 and continuing for 10 days or until neutrophil count is at least 1000/mm3. Treatment continues every 3 weeks for a minimum of 6 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve at least stable response receive GM-CSF 3 times a week for up to 2 years. Patients are followed every 3-6 months.

PROJECTED ACCRUAL: A maximum of 30 patients will be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven multiple myeloma Pancytopenia related to multiple myeloma allowed Failed or progressed after at least 2 chemotherapy or biologic therapy regimens

PATIENT CHARACTERISTICS: Age: 16 and over Performance status: Not specified Life expectancy: Not specified Hematopoietic: Platelet count at least 50,000/mm3 Absolute neutrophil count at least 750/mm3 Hepatic: SGOT/SGPT less than 3 times upper limit of normal Bilirubin less than 5.0 mg/dL Renal: Not specified Other: No active infection requiring intravenous antibiotics Not HIV positive Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics May have failed prior bone marrow transplant No other concurrent colony stimulating factors Concurrent immunoglobulin allowed Chemotherapy: See Disease Characteristics Concurrent pamidronate allowed Endocrine therapy: Not specified Radiotherapy: Concurrent standard radiation therapy to treat extra-skeletal and/or skeletal tumor sites allowed Surgery: Not specified Other: Concurrent epoetin alfa for anemia allowed

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1998-10; Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad A. Hussein, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Cancer Center, Cleveland, Ohio, United States